CLINICAL TRIAL: NCT02518061
Title: Role of 11C-Methionine PET for the Prognostic and Molecular Characterization of Gliomas Candidate to Surgery.
Brief Title: 11C-Methionine PET as Prognostic Marker of Gliomas
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 1418
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Glioma
Keywords: Glioma; 11C-Methionine PET
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Tumor surgical specimen
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — This is a retrospective study

SUMMARY:
This is a retrospective study that involves the revision of clinical, instrumental and pathologic data of an estimated cohort of maximum 145 patients with glioma treated with surgery with radical intent at our center.

DETAILED DESCRIPTION:
This is a retrospective observation that involves the revision of clinical, instrumental and pathologic data of an estimated cohort of 145 patients with glioma treated with surgery with radical intent at our center.

We will review 11C-Methionine PET data acquired within 30 days prior to surgery and analyze its principal imaging characteristics with respect to IDH1 mutation status, MGMT promoter methylation and 1p/19q co-deletion. These markers will be studied on tumor tissue obtained at surgery, used for diagnostic purposes and stored in paraffin.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of glioma
* 11C-Methionine within 30 days before surgery

Exclusion Criteria:

* Absence of tumor specimen
* No clinical data
* 11C-Methionine can not be evaluated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit a maximum number of 145 patients with glioma operated in our institution during 2011-2015, of which are available clinical and instrumental data and surgical tumor specimen.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2015-07; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation of SUVmax (Maximal Standardized Uptake Value) in patients with glioma undergoing surgery with IDH1 mutation, MGMT promoter methylation and 1p/19q co-deletion, | Baseline SUVmax up to 1 month before surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Egesta Lopci, MD, Principal Investigator — Humanitas Clinical and Research Hospital
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopci E, Franzese C, Grimaldi M, Zucali PA, Navarria P, Simonelli M, Bello L, Scorsetti M, Chiti A. Imaging biomarkers in primary brain tumours. Eur J Nucl Med Mol Imaging. 2015 Apr;42(4):597-612. doi: 10.1007/s00259-014-2971-8. Epub 2014 Dec 18. PMID 25520293
- [Background] Schinkelshoek M, Lopci E, Clerici E, Alongi F, Mancosu P, Rodari M, Navarria P, van der Hiel B, Scorsetti M, Chiti A. Impact of 11C-methionine positron emission tomography/computed tomography on radiation therapy planning and prognosis in patients with primary brain tumors. Tumori. 2014 Nov-Dec;100(6):636-44. doi: 10.1700/1778.19268. PMID 25688497
- [Background] Navarria P, Reggiori G, Pessina F, Ascolese AM, Tomatis S, Mancosu P, Lobefalo F, Clerici E, Lopci E, Bizzi A, Grimaldi M, Chiti A, Simonelli M, Santoro A, Bello L, Scorsetti M. Investigation on the role of integrated PET/MRI for target volume definition and radiotherapy planning in patients with high grade glioma. Radiother Oncol. 2014 Sep;112(3):425-9. doi: 10.1016/j.radonc.2014.09.004. Epub 2014 Oct 9. PMID 25308182
- [Background] Riva M, Lopci E, Castellano A, Olivari L, Gallucci M, Pessina F, Fernandes B, Simonelli M, Navarria P, Grimaldi M, Ruda R, Castello A, Rossi M, Alfiero T, Soffietti R, Chiti A, Bello L. Lower Grade Gliomas: Relationships Between Metabolic and Structural Imaging with Grading and Molecular Factors. World Neurosurg. 2019 Jun;126:e270-e280. doi: 10.1016/j.wneu.2019.02.031. Epub 2019 Feb 22. PMID 30797926
- [Background] Lopci E, Riva M, Olivari L, Raneri F, Soffietti R, Piccardo A, Bizzi A, Navarria P, Ascolese AM, Ruda R, Fernandes B, Pessina F, Grimaldi M, Simonelli M, Rossi M, Alfieri T, Zucali PA, Scorsetti M, Bello L, Chiti A. Prognostic value of molecular and imaging biomarkers in patients with supratentorial glioma. Eur J Nucl Med Mol Imaging. 2017 Jul;44(7):1155-1164. doi: 10.1007/s00259-017-3618-3. Epub 2017 Jan 21. PMID 28110346
- [Background] Castello A, Riva M, Fernandes B, Bello L, Lopci E. The role of 11C-methionine PET in patients with negative diffusion-weighted magnetic resonance imaging: correlation with histology and molecular biomarkers in operated gliomas. Nucl Med Commun. 2020 Jul;41(7):696-705. doi: 10.1097/MNM.0000000000001202. PMID 32371671
- [Background] Riva M, Rodriguez Y Baena R, Pessina F, Lopci E, Fernandes B, Galli C, Rossi M, Bello L. The diffusion-weighted imaging and 11-C-methionine positron emission tomography depiction of an endodermal cyst at the cervico-medullary junction. Br J Neurosurg. 2015;29(5):739-41. doi: 10.3109/02688697.2015.1023780. Epub 2015 Mar 26. PMID 25812023